CLINICAL TRIAL: NCT07361185
Title: A Sticker Reminder Intervention to Promote Intravenous-to-Oral Fluoroquinolone Switching: A Cluster-Randomized Controlled Trial
Brief Title: A Sticker Reminder Intervention to Promote IV-to-PO Fluoroquinolone Switching
Acronym: STICKER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 373/2563(IRB1)
Record Dates: First submitted 2026-01-04; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Fluoroquinolone; Adult
Keywords: Antimicrobial stewardship; Fluoroquinolone; Antibiotic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): No AMs intervention
- Sticker reminder arm (Experimental): Sticker reminder
  Interventions: Behavioral: Sticker reminder

INTERVENTIONS:
Behavioral: Sticker reminder — a reminder sticker was applied to the vital signs sheet of patients meeting predefined switching criteria
  Arms: Sticker reminder arm

SUMMARY:
A single-center, cluster-randomized controlled trial was conducted to determine the effect of Sticker reminder intervention on IV-to-PO switching of fluoquinolone.

DETAILED DESCRIPTION:
A single-center, cluster-randomized controlled trial was conducted across 44 general wards at Siriraj Hospital, Thailand, from July 2020 to December 2024. The study population consisted of adult patients who received at least one dose of intravenous fluoroquinolones. Wards were randomized in a 1:1 ratio to either the sticker reminder intervention or standard care. In the intervention group, a reminder sticker was applied to patients' vital signs sheets when predefined IV-to-oral switching criteria were met. The primary outcome was the proportion of intravenous-to-oral fluoroquinolone switching in the intention-to-treat (ITT) and modified intention-to-treat (mITT) populations.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (aged ≥ 18 years)
2. Diagnosis of any infection
3. Receiving at least one dose of intravenous fluoroquinolones (ciprofloxacin, levofloxacin, or moxifloxacin)

Exclusion Criteria:

1. Inability to tolerate oral medications (e.g., due to severe nausea/vomiting, malabsorption, active gastrointestinal bleeding, or severe diarrhea);
2. Being in an immunodeficiency state (e.g., neutropenia [absolute neutrophil count ≤ 500 cells/mm3], symptomatic HIV/AIDS, history of bone marrow or organ transplantation, leukemia, or current use of immunosuppressive agents); or
3. Having severe infections requiring exclusive intravenous antimicrobial therapy (e.g., infective endocarditis, meningitis, encephalitis, brain abscess, or prosthetic device infections).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
IV-to-PO switching | From the day of initiation of fluoroquinolone to the discharge date (Up to 1 year)
  Proportion of patients who underwent switching from intravenous fluoroquinolone to oral fluoroquinolone within the same hospitalization

SECONDARY OUTCOMES:
Length of stay | From the day of initiation of intravenous fluroquinolone to the day of discharge (up to 1 year)
  The total length of hospital stay of that given admission
Duration of FQ therapy | From the first day to the last day of fluroquinolone use (up to 1 year)
  The total duration of intravenous fluroquinolone and oral fluroquinolone (day)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No